CLINICAL TRIAL: NCT07324889
Title: An Open-label, Single-arm, Prospective, Multicenter, Phase I/II Clinical Study on the Safety and Efficacy of CD19/BCMA CAR-T Cell Therapy for Relapsed/Refractory Warm Antibody Autoimmune Hemolytic Anemia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yihao Wang (Other)
Responsible Party: Sponsor-Investigator, Yihao Wang, Associate Chief Physician, Tianjin Medical University General Hospital
Organization: Tianjin Medical University General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2025-YX-220-01
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-10

CONDITIONS: Relapsed/Refractory Warm Antibody Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/BCMA CAR-T Cell Therapy for Relapsed/Refractory Warm Antibody Autoimmune Hemolytic Anemia (Other)
  Interventions: Drug: CD19/BCMA CAR-T

INTERVENTIONS:
Drug: CD19/BCMA CAR-T — Eligible participants should receive preconditioning 5 to 3 days before CAR-T cell infusion. The recommended preconditioning regimen is fludarabine (30 mg/m²/day for 3 consecutive days) and cyclophosphamide (300 mg/m²/day for 3 consecutive days) (Flu/Cy). Thirty minutes before infusion, medications for preventing allergic reactions should be administered: 25 mg of promethazine hydrochloride or 12.5 mg of diphenhydramine, which can be given intramuscularly or orally. Adopting the two-stage optimal design proposed by Bryant and Day, it is planned to enroll 24 subjects with relapsed/refractory warm antibody autoimmune hemolytic anemia, with a selected dosage of 1×10⁶ CAR⁺ cells/kg.

SUMMARY:
This study is an open-label, single-arm, prospective, multicenter, phase I/II clinical trial. It adopts the two-stage optimal design proposed by Bryant and Day to investigate the efficacy, safety, and in vivo pharmacokinetic characteristics of CD19/BCMA CAR-T cell therapy in the treatment of relapsed/refractory warm antibody autoimmune hemolytic anemia.

DETAILED DESCRIPTION:
With reference to the protocol by the team led by Georg Schett from Germany, a dosage of 1×10⁶ CAR⁺ cells per kilogram was selected, and it is planned to enroll 24 subjects with relapsed/refractory warm antibody autoimmune hemolytic anemia (wAIHA).

The two-stage optimal design proposed by Bryant and Day was adopted:

Stage 1: A total of 8 participants will be enrolled, with the core objective of evaluating the tolerance to treatment-related toxicity. By monitoring safety events (including grade ≥2 cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity syndrome (ICANS), and grade 3-4 neutropenia lasting more than 28 days, etc.), it will be determined whether the number of such events is ≤ 5.

Stage 2: A total of 16 participants will be enrolled, focusing on assessing treatment response, which requires that at least 4 participants achieve a definite therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years and ≤ 75 years.
2. Meeting the criteria for relapsed/refractory warm antibody autoimmune hemolytic anemia (wAIHA), and the patient must have received treatment with at least one of rituximab or cyclophosphamide.
3. Criteria for diagnosing relapsed/refractory warm antibody AIHA: It refers to warm antibody AIHA in which the patient has poor response to first-line and second-line or above standard treatments (e.g., glucocorticoids), or the disease recurs after effective treatment, or the patient requires continuous or repeated treatment to control the disease.
4. Disease duration of more than 6 months, with persistent disease activity or progression despite receiving conventional treatment for ≥ 2 months, or recurrence of disease activity after disease remission. Definition of conventional treatment: Use of glucocorticoids plus at least one of the following immunomodulators: cyclophosphamide, cyclosporine, and biological agents (including rituximab, etc.).
5. No systemic active infection (e.g., infectious pneumonia, pulmonary tuberculosis) within 2 weeks before leukapheresis.
6. Expected survival time of more than 3 months from the date of signing the informed consent form.
7. Peripheral blood routine meeting the following requirements simultaneously: absolute neutrophil count (ANC) ≥ 1000/μL; hemoglobin (HGB) ≥ 60 g/L; platelet count (PLT) ≥ 30,000/μL.

   Hepatic, renal, cardiopulmonary functions meeting the following requirements:
   1. Creatinine ≤ 1.5 × upper limit of normal (ULN);
   2. Left ventricular ejection fraction (LVEF) ≥ 50%;
   3. Oxygen saturation > 90%;
   4. Total bilirubin ≤ 4 × ULN;
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN.
8. Studies in patients with an Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
9. Female study participants of childbearing potential (defined as all female participants who are physiologically capable of becoming pregnant) must agree to use highly effective contraceptive methods from at least 28 days before the start of lymphodepletion until 2 years after CAR-T cell infusion (including the period of study treatment with dose interruptions). Male participants whose partners are of childbearing potential must agree to use effective barrier contraceptive methods from the start of lymphodepletion until 2 years after CAR-T cell infusion, and must not donate semen or sperm throughout the study period.
10. Female study participants of childbearing potential must have a negative result in serum beta-human chorionic gonadotropin (β-hCG) testing both at screening and within 48 hours before the first dose of lymphodepletion treatment.
11. Participants must voluntarily agree to participate in this study and sign the informed consent form. Vulnerable populations may be included in the study. If a study participant is unable to read or sign the informed consent form due to incapacity or other reasons, their legal guardian must act as a proxy to go through the informed consent process and sign the form. If a study participant is unable to read the informed consent form (e.g., illiterate participants), a witness must be present to observe the informed consent process and sign the form.

Exclusion Criteria:

1. Concomitant diagnosis of any type of tumor, which is deemed unsuitable for participation in this study by the investigator.
2. A history of clinically significant central nervous system (CNS) diseases or pathological changes caused by non-autoimmune diseases prior to screening, including but not limited to: cerebrovascular accident, aneurysm, epilepsy, convulsions/seizures, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
3. A history of major organ transplantation (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation.
4. Presence of IgA deficiency at screening (serum IgA level < 10 mg/dL).
5. Presence of any of the following conditions at screening:

   1. Active hepatitis (hepatitis B virus deoxyribonucleic acid [HBV-DNA] or hepatitis C virus ribonucleic acid [HCV-RNA] test results above the lower limit of detection);
   2. Human immunodeficiency virus (HIV) infection, known acquired immunodeficiency syndrome (AIDS), or syphilis infection.
6. A history of any of the following cardiovascular diseases within 6 months prior to screening: New York Heart Association (NYHA) Class III or IV heart failure, myocardial infarction, unstable angina pectoris, uncontrolled or symptomatic atrial arrhythmia, any ventricular arrhythmia, or other heart diseases with significant clinical significance.
7. Having received any of the following treatments for autoimmune diseases:a) Use of therapeutic-dose corticosteroids (defined as prednisone or its equivalent > 20 mg/day) within 7 days before leukapheresis;b) Use of any other investigational drugs for autoimmune diseases within 4 weeks before leukapheresis, except for cases where the drug was ineffective or disease progressed during the investigational treatment, and at least 3 half-lives have passed before leukapheresis (enrollment is permitted in such cases);c) Previous receipt of CAR-T cell therapy or other genetically modified T cell therapies.
8. A history of grade ≥ 2 bleeding within 30 days before screening, or long-term continuous treatment with anticoagulant drugs (e.g., warfarin, low-molecular-weight heparin, or factor Xa inhibitors, etc.).
9. Having undergone plasma exchange, plasmapheresis, hemodialysis, or intravenous immunoglobulin (IVIG) administration within 14 days before leukapheresis.
10. Use of any live vaccines for infectious diseases within 8 weeks before CAR-T cell infusion.
11. Pregnant or lactating women.
12. Known life-threatening allergic reactions, hypersensitivity reactions, or intolerance to the CAR-T cell preparation or its excipients (including DMSO).
13. Poor compliance of the study participant as judged by the investigator, or unwillingness or inability to comply with other requirements of the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | Within 28 days after CAR-T infusion
  Evaluate the number of cases, incidence rate, and severity of various adverse events after CD19/BCMA CAR-T infusion, mainly focusing on immunotherapy-related toxic reactions such as cytokine release syndrome (CRS), immune effector cell therapy-associated

SECONDARY OUTCOMES:
Pharmacokinetics-AUC(0~28days) | Day 7, Day10, Day 14, Day 28 after treatment
  Area under the curve of CAR T cells from time zero to Day 28
Overall response rate (ORR) evaluated by the investigators | Day 28, Month 3, Month 6 after treatment
  Efficacy of CD19/BCMA CAR-T in the treatment of refractory autoimmune diseases, include: complete response (CR) rate and partial response (PR) rate (defined as a reduction of ≥50% in disease activity) at day28, month 3 and month 6 after treatment;
Changes in immunological indicators and hemolysis-related indicators after infusion. | Day 28, Month 2, Month 3, Month 6, Month 12, and Month 24 after treatment
  Bilirubin, LDH, conjugated hemoglobin, free hemoglobin, Direct anti human globulin test (DAT) etc
Pharmacokinetics-Tmax | Day 7, Day10, Day 14, Day 28 after treatment
  Time to peak transgene level
Pharmacokinetics-Tlast | Day7, Day10, Day14, Day28, Month2 , Month3 , Month6 , Month9, Month12 after treatment
  The longest detectable CART copy number time (day)
Progression-free Survival (PFS) | Minimum of 1 years post CAR-T infusion
  Time from CAR-T infusion to first documentation of progressive disease (PD), or death due to any cause, whichever occurs first